CLINICAL TRIAL: NCT00743080
Title: GYNAECARE MORCELLEX Tissue Morcellator vs. ROTOCUT GI Tissue Morcellator: a Randomized Controlled Study
Brief Title: Randomized Controlled Trial (RCT)Comparing GYNAECARE MORCELLEX Versus ROTOCUT GI Tissue Morcellators
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Collaborators: Johnson & Johnson (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300-07-015
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2008-08

CONDITIONS: Uterine Myomas
Keywords: laparoscopy; myomectomy; myomas; morcellator; supracervical hysterectomy; surgery; symptomatic uterine myomas
MeSH Terms: conditions — Myoma

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): Laparoscopic myomectomy and supracervical hysterectomy using GYNECARE MORCELLEX
  Interventions: Procedure: Laparoscopic myomectomy and supracervical hysterectomy with GYNECARE MORCELLEX
- 2 (Active Comparator): Laparoscopic myomectomy and supracervical hysterectomy using ROTOCUT G1
  Interventions: Procedure: Laparoscopic myomectomy and supracervical hysterectomy with ROTOCUT G1

INTERVENTIONS:
Procedure: Laparoscopic myomectomy and supracervical hysterectomy with GYNECARE MORCELLEX — Laparoscopic myomectomy with GYNECARE MORCELLEX: Laparoscopic approach. Longitudinal incision close to the midline of myoma. Identification of cleavage plane. Enucleation of myoma. Suturing myometrial. Removal of myoma with a automatic morcellator (GYNECARE MORCELLEX).
  Laparoscopic supracervical hysterectomy using GYNECARE MORCELLEX: Laparoscopic approach. Use of bipolar diathermy and scissor starting with the round ligament and then the utero-ovarian ligament, otherwise the infundibulopelvic ligament in case of removal of adnexa. Identification, desiccation with polar diathermy, and transection of the uterine vessels. Repetition of the procedure on the contra-lateral side. Opening of vagina just below uterine vessels using an unipolar needle. Removal of uterus by means of GYNECARE MORCELLEX. Abdominal cavity irrigation.
  Arms: 1
Procedure: Laparoscopic myomectomy and supracervical hysterectomy with ROTOCUT G1 — Laparoscopic myomectomy with ROTOCUT G1: Laparoscopic approach. Longitudinal incision close to the midline of myoma. Identification of cleavage plane. Enucleation of myoma. Suturing myometrial. Removal of myoma with a automatic morcellator (ROTOCUT G1).
  Laparoscopic supracervical hysterectomy using ROTOCUT G1: Laparoscopic approach. Use of bipolar diathermy and scissor starting with the round ligament and then the utero-ovarian ligament, otherwise the infundibulopelvic ligament in case of removal of adnexa. Identification, desiccation with polar diathermy, and transection of the uterine vessels. Repetition of the procedure on the contra-lateral side. Opening of vagina just below uterine vessels using an unipolar needle. Removal of uterus by means of ROTOCUT G1. Abdominal cavity irrigation.
  Arms: 2

SUMMARY:
To date, laparoscopic approach may apply to several gynecologic diseases. Among the recent advances in laparoscopy an important role was assumed by the methods of tissue extraction. In particular electronic power morcellators have become instruments of large use in surgical practice.

The tissue morcellator is an endoscopic instrument indicated for cutting, coring and extracting tissue in operative laparoscopy, and it has a pivotal role during specific gynaecologic procedures as well as myomectomy and hysterectomy. The main advantages offered by electronic morcellator consist in reduction of operative time and of risk in hernia formation, this last due to the absence of fascia's tearing or stretching.

Recently, a new generation of tissue morcellator has been commercialized. In particular, GYNECARE MORCELLEX (Ethicon-Johnson & Johnson Gateway, US) and ROTOCUT G1 (Karl Storz, Culver City, CA, US) are two tissue morcellators currently available. These instruments seem to offer advantages over the previous models in terms of precision, speed and durability. The most useful of this features seems to be the higher speed, in particular it has been calculated that they morcellate tissues approximately four times faster than those of the previous generation. The high speed that characterizes this new morcellator potentially results in reduced operative time with consequent benefits in other surgical outcomes such as postoperative pain and recovery time.

Even if both morcellator seems to be high-quality instruments, no study was designed until now to compare these two tools in a prospective fashion.

DETAILED DESCRIPTION:
Patients with symptomatic uterine leiomyomas will be assessed for eligibility and will be enrolled in the present protocol-study.

At entry, in each woman age, parity, body mass index (BMI), menopausal, socioeconomic and work status, symptoms related to the gynecologic disease, previous major surgical laparotomies, and associated medical condition will be assessed.

All eligible patients will be randomized in single blocks using a central computer generating randomization lists (University of Catanzaro). The subjects will be assigned to one of four subgroups of surgical treatment, i.e. group A1 myomectomies performed using GYNECARE MORCELLEX, group A2 supracervical hysterectomies performed using GYNECARE MORCELLEX, group B1 myomectomies performed using ROTOCUT G1 and group B2 supracervical hysterectomies performed using ROTOCUT G1.

Before surgery, for each patient gynaecological and rectal examination, Papanicolau smear test, ultrasonographic and hysteroscopic assessment with endometrial biopsy will be performed.

For each surgical intervention the following parameters will be recorded: duration of surgical procedures, intra-operative blood loss, amount of blood transfusion, intra-operative complications, number of laparotomic conversion, postoperative pain, post-operative complications, hospital stay, and time to return to full activity and/or work.

Data will be analyzed using the intention-to-treat principle and a P value of 0.05 or less will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic uterine leiomyomas with main diameter over 5 cm

Exclusion Criteria:

* Major medical conditions
* Endocrinologic diseases
* Current or past, acute or chronic psychiatric disorders
* Premenstrual syndrome
* Use of drugs influencing cognition, vigilance and/or mood within six months of the study enrolment
* Hypoechoic or calcified leiomyomas at ultrasound
* Associated lesions in the uterus and adnexa at ultrasound
* Pattern of hyperplasia with cytologic atypia in the endometrial biopsy
* Abnormal Papanicolau smear test
* Positive urine pregnancy test result

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-01; Study Completion 2010-01

PRIMARY OUTCOMES:
Morcellament time

SECONDARY OUTCOMES:
Total operative time
Feasibility [subjective score of difficulty]
Blood loss
Post-operative complications | 12 months
Postoperative pain
Hospital stay
Time to return to full activity and/or work | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, MD, PhD, Principal Investigator — Department of Experimental and Clinical Medicine, University "Magna Graecia" of Catanzaro, - Viale Europa Loc. Germaneto 88100 Catanzaro, Italy
Locations (1):
- University Magna Graecia, Catanzaro, Italy, Italy

REFERENCES:
- [Result] Zullo F, Falbo A, Iuliano A, Oppedisano R, Sacchinelli A, Annunziata G, Venturella R, Materazzo C, Tolino A, Palomba S. Randomized controlled study comparing the Gynecare Morcellex and Rotocut G1 tissue morcellators. J Minim Invasive Gynecol. 2010 Mar-Apr;17(2):192-9. doi: 10.1016/j.jmig.2009.11.009. PMID 20226407